CLINICAL TRIAL: NCT06209528
Title: Assessing Neurophysiological Function, Cognitive Function, and Health-related Quality of Life in School Children: a Feasibility Study
Brief Title: Assessing Neurophysiological and Cognitive Function in School Children
Acronym: WIS
Status: Completed | Type: Observational
Sponsor: Life University (Other)
Collaborators: New Zealand College of Chiropractic (Unknown)
Responsible Party: Sponsor
Other Study IDs: I-0028
Record Dates: First submitted 2024-01-08; First posted 2024-01-17 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Pediatric ALL
Keywords: pediatrics; EEG; cognition; autonomic nervous system; HRV
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- School-aged children: No intervention

SUMMARY:
This trial will investigate the feasibility of implementing our novel assessment battery in a neurodiverse pediatric population. More specifically, we want to assess our processes and procedures with respect to 1) recruitment rate (i.e., efficiency of our recruitment methods), 2) tolerability (i.e., proportion of participants able to wear the hardware without difficulty), 3) compliance (i.e., proportion of participants able to complete each task as instructed), 4) efficiency (i.e., time to completion of the test battery), and 5) data fidelity (i.e., proportion of test acquisitions with data suitable for subsequent analyses).

DETAILED DESCRIPTION:
The total estimated time requirement for this study is ~60 minutes (i.e., two ~30-minute sessions) and wearing a FitBit for 7 days.

Per their normal and customary procedures, Drs. Amanda and Lona will send a cover letter home to the parent(s)/guardian(s) of their patients introducing the study along with the informed consent (IC) form. Parent(s)/guardian(s) will be asked to indicate their level of interest on the letter and return it (along with the IC, if applicable) to the school. Parents/guardians who indicate that they have additional queries will be contacted by a member of our research staff via the parent's/guardian's preferred method (i.e., phone, text, and/or email). A signed IC will be required prior to enrolling any student in the study.

Up to 20 students (ages 5-17) will be tested over the course of 1 week.

This study will be conducted in designated testing rooms at participating schools within the Chippewa Falls district (Wisconsin, USA). A researcher will sit down with each student and review the age-appropriate informed assent (IA) form. Even if their parent(s)/guardian(s) would like them to participate, students must acknowledge their willingness to participate verbally (e.g., "yes I would like to do the study") and/or physically (e.g., nod their head & give a thumbs up) and sign the IA form to be enrolled in the study.

The primary aims of this trial are to investigate the feasibility of implementing our novel assessment battery with a neurodiverse pediatric population. More specifically, we want to assess our processes and procedures with respect to 1) recruitment rate (i.e., number of subjects recruited within the 1 month recruitment window), 2) tolerability (i.e., proportion of participants able to wear the hardware without difficulty), 3) compliance (i.e., proportion of participants able to complete each task as instructed), 4) efficiency (i.e., time to completion of the test battery), and 5) data fidelity (i.e., proportion of test acquisitions with data suitable for subsequent analyses). This feasibility trial is intended inform a future cluster randomized controlled trial (RCT) assessing the effects of chiropractic care on a neurodiverse pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* 5-17 years old
* Student of the Chippewa Falls school district
* Parent(s)/Guardian(s) provide signed informed consent
* Child able to provide signed informed assent & acknowledge desire to participate verbally (e.g., "Yes, I want to do the study") and/or physically (e.g., nods head & gives thumbs up).

Exclusion Criteria:

* Unable to perform assessments due to movement limitations (e.g., confined to a wheelchair)
* Unable to perform the assessments due to contraindications (e.g., has a disorder that causes fainting during postural changes such as POTS or orthostatic hypotension)
* Pacemaker or known heart condition that influences the electrical function of the heart
* Deemed to be at "high risk" of suicide per the C-SSRS

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: School-age children
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Recruitment period (1 week)
  Total number of subjects enrolled
Protocol tolerability | Study period (2 school weeks)
  Proportion of participants able to tolerate wearing a given piece of acquisition hardware (i.e., EEG cap, ECG sensors, FitBit) for the duration of the study period
Participant compliance | Study period (2 school weeks)
  Proportion of participants able to comply with the instructions for a given task
Protocol efficiency | 1 school week
  Average time to completion for both of the 1-day assessment sessions
Data fidelity | Study period (2 school weeks)
  Proportion of acquisitions for a given task with data suitable for subsequent analysis

CONTACTS AND LOCATIONS:
Overall Officials: Tyson Perez, PhD, Principal Investigator — Life University
Locations (1):
- Chippewa Falls Area Unified School District, Chippewa Falls, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No